CLINICAL TRIAL: NCT00274313
Title: A Study of the Safety and Pharmacokinetics of 552-02 Following 14 Days of Dosing By Inhalation in Patients With Cystic Fibrosis
Brief Title: Safety Study of Inhaled 552-02 in Cystic Fibrosis Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Parion Sciences (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Parion 552-203
Record Dates: First submitted 2006-01-06; First posted 2006-01-10 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

INTERVENTIONS:
Drug: 552-02

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of a new inhaled sodium-channel blocker called 552-02 in teens and adults with cystic fibrosis. 552-02 will be inhaled once a day for 14 days using a nebulizer. A small subgroup of patients will donate blood samples for pharmacokinetic analysis to see how 552-02 is absorbed into the blood and eliminated after 14 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged > 14 years.
2. Patients who are diagnosed with cystic fibrosis.
3. Patients who have a FEV1 ≥ 50% predicted (post-bronchodilator) at screening.
4. Patients who are able to perform reproducible spirometry according to ATS guidelines.
5. Patients who have an oxygen saturation of ≥ 92% on room air as determined by pulse oximetry at screening.

Exclusion Criteria:

1. Patients who have a FEV1 change ≥ 15% after bronchodilator use at screening.
2. Patients who have unstable lung disease as defined by the requirement for intravenous antibiotics during the four weeks prior to screening, a change in medical regimen within 14 days prior to administration of the first dose of study drug or during the 14 day treatment period, a FEV1 ≥ 15% below recent (within six months) clinical measurements, or significant new findings on chest radiograph (pneumothorax, lobar/segmental collapse) that are not considered a part of the usual, chronic progression of cystic fibrosis lung disease.
3. Patients on angiotensin converting enzyme (ACE) inhibitors.
4. Patients with renal insufficiency as evidenced by hyperkalemia (blood potassium levels greater than 5.5 mEq/L) or serum creatinine > 2.0 mg/dL.
5. Patients who have a history of drug allergies to any medicine chemically related to the study drug (e.g. amiloride, Moduretic, Midamor; triamterene).
6. Patients who are pregnant, have a positive pregnancy test, or are nursing.
7. Patients who have had a lung transplant.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2006-01; Study Completion 2006-08

PRIMARY OUTCOMES:
Safety assessments
Blood and urine laboratory tests
Pulmonary function tests
Electrocardiograms
Vital signs and pulse oximetry

SECONDARY OUTCOMES:
Plasma pharmacokinetics on Day 14 of the study.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - University of California at San Diego, San Diego, California
  - University of California at San Francisco Medical Center, San Francisco, California
  - The Children's Hospital, Denver, Colorado
  - Nemours Children's Clinic, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Children's Memorial Hospital, Chicago, Illinois
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Morristown Memorial Hospital, Morristown, New Jersey
  - State University of New York Upstate, Syracuse, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Virginia, Charlottesville, Virginia